CLINICAL TRIAL: NCT06501170
Title: Risk Factors of Adverse Outcomes After Emergency Abdominal Emergency Surgery and Establishment of a Risk Stratification Tool
Brief Title: Risk Stratification for Abdominal Emergency Surgery: a Cohort Study
Status: Active, not recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K6243
Record Dates: First submitted 2024-06-26; First posted 2024-07-15 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Emergency Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Retrospective Data Analysis of Emergency Abdominal Surgery Outcomes — Retrospective Data Analysis of Emergency Abdominal Surgery Outcomes

SUMMARY:
The goal of this retrospective observational study is to identify risk factors of unwanted outcomes (in-hospital morbidity and mortality) among patients undergoing emergency abdominal surgery.

DETAILED DESCRIPTION:
Patients undergoing emergency abdominal surgery at a single tertiary care institution with a high volume of emergency abdominal surgeries, especially for high-acuity patients, between January 1, 2023, and June 1, 2024, will be included. Baseline demographics, indication for surgery, and preoperative status (respiratory support, cardiovascular stability, Glasgow score, SOFA score, preoperative lab results, and preoperative waiting time including Time to Theatre (TTT) and Time to Knife (TTK)) will be recorded.

Definitions:

Time to Theatre (TTT): The duration from when it is determined that the patient needs surgery to the time the patient arrives at the operating theatre.

Time to Knife (TTK): The duration from when the patient enters the operating theatre to the time the first incision is made.

These data will be retrieved from the electronic health record system.

Intraoperative factors, including ASA classification, anesthesia method, type of surgical intervention, intraoperative lab results, transfusions, input/output (I/O), inotropic/vasopressor usage, and discharge ward, will also be retrieved from the electronic health record system. Postoperative outcomes, including in-hospital mortality and morbidity (complications stratified by the Clavien-Dindo classification system), will be assessed by trained investigators. Secondary outcomes include postoperative length of hospital stay and health care costs.

A statistical model will be built to identify risk factors for morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing emergency abdominal surgery at a single tertiary care institution between January 1, 2023, and June 1, 2024

Exclusion Criteria:

Repeated surgery for the same patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing emergency abdominal surgery at a single tertiary care institution between January 1, 2023, and June 1, 2024.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
in-hospital mortality | From date of surgery until discharge day, assessed up to 4 weeks
  documented in-hospital mortality
in-hospital morbidity | From date of surgery until discharge day, assessed up to 4 weeks
  in-hospital postoperative complications classified using Clavein-Dindo score

SECONDARY OUTCOMES:
postoperative length of hospital stay | From date of surgery until discharge day, assessed up to 4 weeks
  postoperative length of hospital stay assessed by days
Health care costs | From date of admission until discharge day, assessed up to 4 weeks
  Health care costs in RMB assessed using hospital billing records

CONTACTS AND LOCATIONS:
Locations (1):
- Lu Che, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No